CLINICAL TRIAL: NCT00033202
Title: Phase I Study of Oral ST1481 Administered Once Weekly Every 3 Out 4 Weeks in Patients With Advanced Solid Malignancies.
Brief Title: This is an Early Study to Investigate the Effect of Gimatecan® in Adults With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sigma-Tau Research, Inc. (Industry)
Collaborators: Rhode Island Hospital (Other); Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST 01-401
Record Dates: First submitted 2002-04-09; First posted 2002-04-10 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Solid Malignancies
Keywords: Solid Tumor; Camptothecin; Pharmacokinetics
MeSH Terms: interventions — ST 1481

INTERVENTIONS:
Drug: Gimatecan® (ST-1481)

SUMMARY:
Gimatecan® is sigma-tau Research's new, potent, oral Topoisomerase I inhibitor. Drugs in this class play a crucial role in destroying DNA replication in tumors. We are conducting this study to determine the Maximum Tolerated Dose of our compound, when given as a capsule, rather than by intravenous injection.

ELIGIBILITY:
Inclusion criteria:

* Histologically/cytologically proven advanced solid tumors
* Life expectancy of at least 3 months with normal hematological, liver and renal function

Exclusion criteria:

* Pregnant and lactating patients
* Participation in any investigating drug study within 4 weeks preceding treatment start or concurrent treatment with any other anti-cancer therapy
* Gastrointestinal dysfunction that could alter absorption or motility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-03; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island